CLINICAL TRIAL: NCT05262569
Title: Increased Postoperative Opioid Use is a Risk Factor for an Ileus After Laparoscopic Colorectal Surgery---A Case Control Study
Brief Title: Postoperative Opioid Use and Ileus Occurrence---A Case Control Study
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Juhui, Assistant professor, Peking University People's Hospital
Other Study IDs: Opioid and postoperative POI
Record Dates: First submitted 2022-02-22; First posted 2022-03-02 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Ileus; Opioid Use
Keywords: ileus; opioid use; enhanced recovery after surgery; colorectal surgery
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ileus group: Patients developed postoperative ileus
  Interventions: Other: ileus
- control group: Patients did not develop postoperative ileus

INTERVENTIONS:
Other: ileus — retrospectively allocation according to a postoperative outcome-ileus
  Groups: ileus group

SUMMARY:
Postoperative ileus (POI) is a significant complication after colorectal surgery, with reported incidence ranging from 10~30%, leading to increased morbidity, hospital length of stay, and thus medical cost. To determine the risk factors for POI is one of the key elements for Enhanced Recovery after Surgery protocol. Increased perioperative opioid usage has been proposed as an independent risk factor for postoperative ileus, as perioperative opioid minimization has proposed to be an effective measure to decrease the incidence of POI. Although opioids are widely used to attenuate stress during surgery, and represent the cornerstone of pain treatment, anesthesiologists are strive to minimize opioid use to decrease opioid-related GI side effects. In this study, the investigators aim to find out the general occurrence of POI in the laparoscopic colorectal surgery and the effects of the postoperative opioid usage on this outcome. The strategies of opioid minimization was also investigated.

DETAILED DESCRIPTION:
2.1 Study design For this case-control study, all elective laparoscopic colorectal procedures performed at a university hospital between Jan 2018 and June 2020 were retrospectively collected by reviewing the institutional colorectal surgery database. The study protocol was approved by the Institutional Review Board of Peking University People's Hospital (2021PHB144-001, May 24, 2021), Beijing, China, and informed consent was waived due to the retrospective design.

The anesthesia medical information system was searched for patients aged 18 years old and above, undergoing elective laparoscopic colorectal procedures who received patient controlled intravenous analgesia postoperatively. Patients were excluded if they had chronic opioid use, converted to open, admitted to intensive care unit(ICU), patient controlled analgesia (PCA) regimens other than sufentanil, PCA used shorter than 48 hours, or incomplete postoperative opioid usage record. Patients were followed up until discharge from the hospital.

2.2 Patient allocation Patients who experienced postoperative ileus were included in ileus group. In accordance with the definition of Vather et al, diagnosis of postoperative ileus required 2 or more of following persistent symptoms on the fourth postoperative day and onward: nausea and vomiting, inability to tolerate solid or semi-liquid diet or failure to pass gas or stool during a 24 hour period, abdominal distension and radiological evidence of ileus. Patient charts, including radiographs were evaluated retrospectively. Diagnosis of an ileus was confirmed clinically and radiographically in all cases. The control group (at a 1:1 ratio) was matched by selecting the same range of age (±5 years of age), the same grade of American Society of Anesthesiology(ASA) classification, and the same types of surgery (colectomy, rectectomy, whole colon resection, or others).

2.3 Perioperative management All patients received standard anesthesia protocol for laparoscopic colorectal procedures within Peking University People's Hospital. Patients might received bilateral transversus abdominis plane(TAP) blocks (0.3% Ropivacaine of 30~40ml under the ultrasound guidance) at the discretion of the anesthesiologist in charge.

General anesthesia was induced using etomidate (0.2-0.6 mg/kg) and sufentanil (0.3 μg/kg) and maintained with continuous infusion of propofol (4-6 mg/kg/h) to target a bispectral index of 40-60. Cisatracurium (0.15 mg/kg) was injected intravenously to facilitate endotracheal intubation. Intravenous sufentanil (0.1 μg/kg) was added before skin incision. During surgery, continuous infusion of remifentanil (0.1-0.2 μg /kg/min) was adjusted to keep heart rate (HR) and mean arterial blood pressure (MAP) within 80-120% of baseline. Hypotension (MAP < 80% of baseline) lasting for 3 min was managed with a bolus of 6 mg of ephedrine or 50 μg of phenylephrine. Bradycardia (HR < 45/min) was treated with atropine (0.25-0.5 mg). At the end of surgery, neostigmine (1 mg) and atropine (0.5 mg) were used to antagonize neuromuscular blockade, and tracheal extubation was performed when the patient was fully awake and breathing adequately. Patients were transferred to the post-anesthesia care unit (PACU) and discharged when the Modified Aldrete Score reached 10.

2.4 Postoperative pain management Postoperative pain management was charged by the acute pain service(APS). Acute pain or side effects related to the opioid was managed through the setting of intravenous patient-controlled analgesia(PCA) device. Patients received intravenous, intramuscular or oral analgesic rescue only after the PCA withdrawal.

In general, a patient-controlled analgesia (PCA) device was attached after tracheal extubation. The PCA was set to provide a bolus of 2~3μg sufentanil (1 μg/ml) with a lockout time of 10~15 min with or without basal infusion, 2~3ml/h (sufentanil 1μg/ml), which was set at the discretion of the anesthesiologist in charge according to the patient's age and weight. After surgery, pain score was verbally rated using the 11-point numeric rating scale (NRS), on which 0 indicates no pain and 10 indicates worst imaginable pain. Patients could self-administer intravenous sufentanil bolus via PCA (2~3μg, 1 μg/ml) postoperatively as rescue analgesia when the NRS score was ≥4, or as needed. PCA was maintained for at least the first 48 h after surgery.

2.5 Study outcomes and measurements Multiple potential risk factors for POI were considered based on literature review. Baseline factors included age(matched), gender, BMI, presence of major comorbidities (cardiovascular diseases, cerebral diseases, pulmonary diseases, or diabetes), ASA classification (matched), and previous abdominal surgery. Operative factors included type of surgery(matched), length of the surgery, estimated blood loss, total input, time to pass stool in patients' without enterostomy, time to tolerance of oral diet, and postoperative length of hospital stay. Analgesia related risk factors included TAP block, intra-operative opioid use(converted into equivalent doses of morphine, mg/kg), postoperative day 1 (POD1) and total post-operative opioid (Sufentanil, μg/kg), and PCA setting (with or without basal infusion). Postoperative NRS at rest and when coughing were recorded. Adverse events occurring prior to discharge were also collected from the hospital chart.

2.6 Statistical analysis Statistical analysis was performed using the SPSS statistical software package (SPSS Inc., Chicago, IL). Continuous variables are expressed as mean ± standard deviation(SD) or medians with interquartile range and categorical variables as numbers and percentages. Between-group differences were evaluated using the independent t test or Mann-Whitney U test for continuous variables and the χ2 test or Fisher exact test for categorical variables, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old and above
* Underwent elective laparoscopic colorectal procedures
* Received patient controlled intravenous analgesia postoperatively

Exclusion Criteria:

* Chronic opioid use
* Converted to open
* Admitted to ICU
* PCA regimens other than sufentanil
* PCA used shorter than 48 hours
* Incomplete postoperative opioid usage record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All elective laparoscopic colorectal procedures performed at a university hospital between Jan 2018 and June 2020 were retrospectively collected by reviewing the institutional colorectal surgery database.
Sampling Method: Probability Sample
Enrollment: 596 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
postoperative opioid usage | Within 3 postoperative days
  Sufentanil(μg/kg) used through patient-controlled analgesia

SECONDARY OUTCOMES:
Use of transversus abdominis plane(TAP) block | Before surgery
  The percentage TAP block of each group
Patent-controlled analgesia(PCA) setting | Within 3 postoperative days
  The percentage of PCA setting with basal infusion

CONTACTS AND LOCATIONS:
Overall Officials: Juhui, Dr., Principal Investigator — Peking University People's Hospital, Beijing, China
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
It need to be discussed within the study group when the results are clear.

REFERENCES:
- [Background] Wu CL, King AB, Geiger TM, Grant MC, Grocott MPW, Gupta R, Hah JM, Miller TE, Shaw AD, Gan TJ, Thacker JKM, Mythen MG, McEvoy MD; Fourth Perioperative Quality Initiative Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Perioperative Opioid Minimization in Opioid-Naive Patients. Anesth Analg. 2019 Aug;129(2):567-577. doi: 10.1213/ANE.0000000000004194. PMID 31082966
- [Background] Artinyan A, Nunoo-Mensah JW, Balasubramaniam S, Gauderman J, Essani R, Gonzalez-Ruiz C, Kaiser AM, Beart RW Jr. Prolonged postoperative ileus-definition, risk factors, and predictors after surgery. World J Surg. 2008 Jul;32(7):1495-500. doi: 10.1007/s00268-008-9491-2. PMID 18305994
- [Background] Pappagallo M. Incidence, prevalence, and management of opioid bowel dysfunction. Am J Surg. 2001 Nov;182(5A Suppl):11S-18S. doi: 10.1016/s0002-9610(01)00782-6. PMID 11755892
- [Background] Camilleri M. Opioid-induced constipation: challenges and therapeutic opportunities. Am J Gastroenterol. 2011 May;106(5):835-42; quiz 843. doi: 10.1038/ajg.2011.30. Epub 2011 Feb 22. PMID 21343919
- [Background] Ahn JH, Ahn HJ. Effect of thoracic epidural analgesia on recovery of bowel function after major upper abdominal surgery. J Clin Anesth. 2016 Nov;34:247-52. doi: 10.1016/j.jclinane.2016.04.042. Epub 2016 May 13. PMID 27687384
- [Background] Stokes AL, Adhikary SD, Quintili A, Puleo FJ, Choi CS, Hollenbeak CS, Messaris E. Liposomal Bupivacaine Use in Transversus Abdominis Plane Blocks Reduces Pain and Postoperative Intravenous Opioid Requirement After Colorectal Surgery. Dis Colon Rectum. 2017 Feb;60(2):170-177. doi: 10.1097/DCR.0000000000000747. PMID 28059913
- [Background] Fields AC, Weiner SG, Maldonado LJ, Cavallaro PM, Melnitchouk N, Goldberg J, Stopfkuchen-Evans MF, Baker O, Bordeianou LG, Bleday R. Implementation of liposomal bupivacaine transversus abdominis plane blocks into the colorectal enhanced recovery after surgery protocol: a natural experiment. Int J Colorectal Dis. 2020 Jan;35(1):133-138. doi: 10.1007/s00384-019-03457-1. Epub 2019 Dec 4. PMID 31797098
- [Background] Pedrazzani C, Menestrina N, Moro M, Brazzo G, Mantovani G, Polati E, Guglielmi A. Local wound infiltration plus transversus abdominis plane (TAP) block versus local wound infiltration in laparoscopic colorectal surgery and ERAS program. Surg Endosc. 2016 Nov;30(11):5117-5125. doi: 10.1007/s00464-016-4862-5. Epub 2016 Mar 22. PMID 27005290
- [Background] Chen JY, Ko TL, Wen YR, Wu SC, Chou YH, Yien HW, Kuo CD. Opioid-sparing effects of ketorolac and its correlation with the recovery of postoperative bowel function in colorectal surgery patients: a prospective randomized double-blinded study. Clin J Pain. 2009 Jul-Aug;25(6):485-9. doi: 10.1097/AJP.0b013e31819a506b. PMID 19542795
- [Background] Aryaie AH, Lalezari S, Sergent WK, Puckett Y, Juergens C, Ratermann C, Ogg C. Decreased opioid consumption and enhance recovery with the addition of IV Acetaminophen in colorectal patients: a prospective, multi-institutional, randomized, double-blinded, placebo-controlled study (DOCIVA study). Surg Endosc. 2018 Aug;32(8):3432-3438. doi: 10.1007/s00464-018-6062-y. Epub 2018 Jan 19. PMID 29352454
- [Background] Jung H, Lee KH, Jeong Y, Lee KH, Yoon S, Kim WH, Lee HJ. Effect of Fentanyl-Based Intravenous Patient-Controlled Analgesia with and without Basal Infusion on Postoperative Opioid Consumption and Opioid-Related Side Effects: A Retrospective Cohort Study. J Pain Res. 2020 Nov 24;13:3095-3106. doi: 10.2147/JPR.S281041. eCollection 2020. PMID 33262644
- [Background] Vather R, Josephson R, Jaung R, Robertson J, Bissett I. Development of a risk stratification system for the occurrence of prolonged postoperative ileus after colorectal surgery: a prospective risk factor analysis. Surgery. 2015 Apr;157(4):764-73. doi: 10.1016/j.surg.2014.12.005. Epub 2015 Feb 25. PMID 25724094
- [Background] Vather R, Bissett IP. Risk factors for the development of prolonged post-operative ileus following elective colorectal surgery. Int J Colorectal Dis. 2013 Oct;28(10):1385-91. doi: 10.1007/s00384-013-1704-y. Epub 2013 May 21. PMID 23689489
- [Background] Grass F, Slieker J, Jurt J, Kummer A, Sola J, Hahnloser D, Demartines N, Hubner M. Postoperative ileus in an enhanced recovery pathway-a retrospective cohort study. Int J Colorectal Dis. 2017 May;32(5):675-681. doi: 10.1007/s00384-017-2789-5. Epub 2017 Mar 11. PMID 28285365
- [Background] Yuan L, O'Grady G, Milne T, Jaung R, Vather R, Bissett IP. Prospective comparison of return of bowel function after left versus right colectomy. ANZ J Surg. 2018 Apr;88(4):E242-E247. doi: 10.1111/ans.13823. Epub 2016 Nov 2. PMID 27806440
- [Background] Kim IK, Kang J, Baik SH, Lee KY, Kim NK, Sohn SK. Impact of prior abdominal surgery on postoperative prolonged ileus after ileostomy repair. Asian J Surg. 2018 Jan;41(1):86-91. doi: 10.1016/j.asjsur.2016.07.006. Epub 2016 Aug 17. PMID 27542335
- [Background] Walter CJ, Maxwell-Armstrong C, Pinkney TD, Conaghan PJ, Bedforth N, Gornall CB, Acheson AG. A randomised controlled trial of the efficacy of ultrasound-guided transversus abdominis plane (TAP) block in laparoscopic colorectal surgery. Surg Endosc. 2013 Jul;27(7):2366-72. doi: 10.1007/s00464-013-2791-0. Epub 2013 Feb 7. PMID 23389068
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Zhen L, Li X, Gao X, Wei H, Lei X. Dose determination of sufentanil for intravenous patient-controlled analgesia with background infusion in abdominal surgeries: A random study. PLoS One. 2018 Oct 17;13(10):e0205959. doi: 10.1371/journal.pone.0205959. eCollection 2018. PMID 30332482
- [Derived] Ju H, Shen K, Li J, Feng Y. Total postoperative opioid dose is an independent risk factor for prolonged postoperative ileus after laparoscopic colorectal surgery: a case-control study. Korean J Anesthesiol. 2024 Feb;77(1):133-138. doi: 10.4097/kja.22792. Epub 2023 Apr 25. PMID 37096402